CLINICAL TRIAL: NCT02604498
Title: Pharmacokinetics Study of Nemonoxacin Malate Capsules in Subjects With Moderate Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Medicine Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: XCNN-150830-1
Record Dates: First submitted 2015-11-03; First posted 2015-11-13 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases | interventions — nemonoxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liver function impaired (Experimental): Subject with Moderate Impaired Hepatic Function. Nemonoxacin Malate Capsules 500mg single dose oral.
  Interventions: Drug: Nemonoxacin
- Healthy Subjects (Experimental): Healthy volunteers. Nemonoxacin Malate Capsules 500mg single dose oral.
  Interventions: Drug: Nemonoxacin

INTERVENTIONS:
Drug: Nemonoxacin — Single dose 500mg oral
  Other Names: Nemonoxacin Malate Capsules

SUMMARY:
This is a single center, open-label, non-randomized, 1:1 parallel control and single dose administration study design. Healthy subjects will be matched to moderate hepatic function impaired (Child-Pugh B，7-9) subjects in age, gender and weight as parallel control, which matches healthy with normal hepatic function according to the of subjects with impaired hepatic function as, after enrollment of subjects with moderate impaired hepatic function (Child-Pugh B，7-9). Hepatic function impaired group and control group both receive orally single-dose of nemonoxacin malate capsule (0.5g). Collect the blood and urine samples before and after the administration to perform pharmacokinetic analysis and safety observation.

DETAILED DESCRIPTION:
Single dose study: evaluate safety and tolerability of oral nemonoxacin capsule 500mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hepatic impairment

  1. male or female aged 18 to 70 years；
  2. has a body mass index of 17 to 30 kg/m2；
  3. eGRF>50ml/min/1.73m2；
  4. Patients in stable condition with moderate impaired hepatic function, due to viral hepatitis, alcoholic liver disease, autoimmune hepatitis, primary biliary cirrhosis or other causes, and determined to be level B according to Child-Pugh classification；
  5. B-ultrasonography, CT or MRI shows or biopsy confirm that have a positive diagnosis of cirrhosis ；
  6. Has stable regimen of treatment of hepatic function impaired for 3 months prior to enrollment;
  7. Female volunteers must meet:

     1. Has sterilization operation, or who are postmenopausal must have been postmenopausal for >1 year, or
     2. Has childbearing potential, but meet the requirement as following:

     Negative pregnancy test prior to enrollment, and Agree with use 1 medical accepted methods of birth control (eg. Hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) during the whole study and continuing until 1 month after the end of the study, and Non-breastfeeding;
  8. Male volunteers must agree to use medical accepted method of birth control (e.g. barrier contraceptive or sexual partner use the method as (7) above) during the study and through 1month after the end of study；
  9. Agree stay in ward prior to dosing within 48h, and agree not to take coffee, tea, chocolate, alcohol, grapefruit juice, orange juice and other food and drink which contain caffeine and xanthine；
  10. Can sign informed consent form on his own accord；
  11. Can comply with study procedures

Healthy subjects without hepatic impairment

1. Male or female volunteers (matched to a subject with hepatic impairment in gender）；
2. Aged 18 to 70 years (matched to a subject with hepatic impairment±5 years, matched range cannot exceed±5 years)；
3. Has a body mass index of 17 to 30 kg/m2（matched to a subject with hepatic impairment±15%，matched range cannot exceed±15%）；
4. Must be in good health as determined by screening medical history, physical examination, vital signs, laboratory test, B ultrasonography and chest X ray；
5. Female volunteers must meet:

   1. Has sterilization operation, or who are postmenopausal must have been postmenopausal for >1 year, or
   2. Has childbearing potential, but meet the requirement as following:

   Negative pregnancy test prior to enrollment, and Agree with use 1 medical accepted methods of birth control (eg. Hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) during the whole study and continuing until 1month after the end of the study, and Non-breastfeeding；
6. Male volunteers must agree to use medical accepted method of birth control (e.g. barrier contraceptive or sexual partner use the method as (7) above) during the study and through 1month after the end of study；
7. Agree stay in ward prior to dosing within 48h, and agree not to take coffee, tea, chocolate, alcohol, grapefruit juice, orange juice and other food and drink which contain caffeine and xanthine；
8. Can sign informed consent form on his own accord；
9. Can comply with study procedures

Exclusion Criteria:

* Subjects with hepatic impairment

  1. Has known or suspected allergies to quinolones, fluoroquinolones, Nemonoxacin or excipients or allergic constitution；
  2. Has acute disease or chronic disease which may affect PK profile of drug in vivo except the disease caused hepatic function impaired；
  3. Has abnormal result of laboratory tests with clinical significance except which caused by the disease of hepatic function impaired；
  4. Has history of clinically significant cardiovascular, neurological or psychiatric, gastrointestinal, pulmonary, renal, endocrine disease prior to study within 1 year；
  5. Has disease seriously affect the immune system such as hematological disease, malignant tumor, or taking immunosuppressant；
  6. Has acute or sub-acute hepatic function failure；
  7. Has experienced esophageal variceal bleeding within the past 6 months；
  8. Has advanced ascites or spontaneous bacterial peritonitis；
  9. Has a history of Gilbert's disease；
  10. Has resistance or liver function abnormal after orally taking nucleoside analogue, an antiviral drug；
  11. Stop taking nucleoside analogue, an antiviral drug within 1 year；
  12. Has total bilirubin>3×upper limit of normal (ULN) and without cholestasis; alkaline phosphatase (ALP)>2×ULN；
  13. Alanine Aminotransferase (ALT)or Aspartate Aminotransferase（AST）>5×ULN；
  14. ALT or AST>3×ULN with total bilirubin>2×ULN；
  15. international senstibity index，INR≥1.5 or prothrombin time activity≤40%；
  16. Child-Pugh assessed as C level；
  17. Has a history of alcoholism within 2 years prior to dosing; drink≥12 times within 3 months prior dosing; alcohol test positive as screening；
  18. Has history of drug misuse within 2 years prior to dosing; urine drug screen positive；
  19. Has history of taking products of tobacco or nicotine more than 5 cigarettes/day within 1 month prior to dosing, or cannot stop smoking during the study;
  20. Use of another investigational drug or drug which can damage hepatic function within 3 months prior to dosing；
  21. Use of drugs affect function of liver metabolism enzyme (e.g. benzene, isopropyl amine, the barbiturates benzodiazepines, marijuana, cocaine, opiates and phencyclidine) within 30 days prior to dosing ；
  22. Has to take the drug which may affect the PK profile of investigate drug (e.g. antacids, sucralfate, metal cation, calcium supplements, warfarin, non-steroidal anti-inflammatory drugs, theophylline, cyclosporine, probenecid and cimetidine) ；
  23. Has gastrointestinal disease or malabsorption syndrome affecting drug Absorb；
  24. Has history of seizures or central nervous system disease which the investigator considers to interfere with compliancy of protocol; or has risk of suicide；
  25. Clinical significant abnormal 12-lead electrocardiograms (ECGs) at screening (eg. atrioventricular block, torsades de pointes ventricular tachycardia (TdT), and other types of ventricular tachycardia, ventricular fibrillation, ventricular flutter, T wave change with clinical significance or any abnormal results of 12-lead ECG which affect QTc interphase) ；
  26. HIV or syphilis RPR test positive；
  27. Conditions investigator consider not suitable to be enrolled in the study. Healthy subjects without hepatic impairment

  <!-- -->

  1. Has known or suspected allergies to quinolones, fluoroquinolones, nemonoxacin or excipients or allergic constitution；
  2. Has a history of alcoholism within 2 years prior to dosing; drink≥12 times within 3 months prior dosing; alcohol test positive as screening；
  3. Has history of drug misuse within 2 years prior to dosing; urine drug screen positive；
  4. Has history of taking products of tobacco or nicotine more than 5 cigarettes/day within 1 month prior to dosing, or cannot stop smoking during the study；
  5. Donated blood or use of another investigational drug within 3 months prior to dosing；
  6. Has history of chronic liver, renal, cardiovascular, neurological or psychiatric, gastrointestinal, pulmonary, urinary, endocrine disease cannot controlled by drugs；
  7. Use of drugs affect function of liver metabolism enzyme within 30 days prior to dosing; or need to take medications which may affect the PK profile of investigational drug (including: products containing Calcium, aluminum, magnesium, iron and zinc, sucralfate, antacid, nutrition supplements, Vitamins and metal supplements) during the study；
  8. Is taking any antibacterial agents or prophylaxis or treatment drugs；
  9. HIV-Ab, HBsAg ,HCV-Ab or syphilis RPR positive；
  10. Clinical significant abnormal 12-lead electrocardiograms (ECGs) at screening (eg. atrioventricular block, torsades de pointes ventricular tachycardia (TdT), and other types of ventricular tachycardia, ventricular fibrillation, ventricular flutter, T wave change with clinical significance or QTc>450ms) ；
  11. Has abnormal result of laboratory test with clinical significance assessed by investigator at screening；
  12. Has gastrointestinal disease or malabsorption syndrome affecting drug Absorb；
  13. Has history of seizures or central nervous system disease which the investigator considers to interfere with compliancy of protocol; or has risk of suicide；
  14. Has any antibacterials, glucocorticoids, immunosuppressive agents or drug may damage organs within 14 days prior to dosing；
  15. Cannot orally take drug；
  16. Has history of or currently has disease and condition may affect the safety and efficancy assessment of investigational drug judged by investigator；
  17. Is a member of the clinical site personnel directly affiliated with this study；
  18. Conditions investigator consider not suitable to be enrolled in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: maximum plasma drug concentration ( Cmax) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: time at which maximum plasma concentration is observed (Tmax) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: area under the plasma concentration vs. time curve (AUC0-t and AUC0-∞) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function:elimination half-life (t1/2) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function:mean dissolution time (MRT) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: total clearance of the drug from plasma (CLz/F) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: Apparent Volume of Distribution (Vz/F) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: cumulative amount of unchanged drug excreted into the urine (Ae Urine 0-24h,0-72h） | Within 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function:renal clearance of the drug from plasma (CLr) | Within 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in Moderate Impaired Hepatic Function: minimum plasma drug concentration (Cmin) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing

SECONDARY OUTCOMES:
Safety assessed by AEs | up to 72 hours after study drug dosing
  reported spontaneously or not by leading questions
Safety assessed by vital signs | up to 72 hours after study drug dosing
  blood pressure, pulse rate, respiratory rate and body temperature
Safety assessed by laboratory tests | up to 72 hours after study drug dosing
  Hematology, blood biochemistry,cogulation test and urinalysis
Safety assessed by physical examination | up to 72 hours after study drug dosing
  (1) general appearance (2) skin (3) head and neck (4)chest, including heart, pulmonary and breast (5) abdomen, including stomach and intestines, liver and gallbladder (6) back (7) Urinary tract (8) extremity (9) neurological or psychiatric system (10) lymph gland (11)others.
Safety assessed by 12-lead ECGs | up to 72 hours after study drug dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Kang Y, Li Y, Xu F, Zhang J, Wang K, Chen Y, Wu J, Guo B, Yu J, Zhang Y. Population Pharmacokinetics Study of Nemonoxacin Among Chinese Patients With Moderate Hepatic Impairment. Clin Ther. 2019 Mar;41(3):505-517.e0. doi: 10.1016/j.clinthera.2019.01.015. Epub 2019 Feb 26. PMID 30819510